CLINICAL TRIAL: NCT06871202
Title: Influence of Manual Therapy on Physical-sport Performance
Brief Title: Manual Therapy and Physical-sport Performance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Juan Elicio Hernández Xumet, PhD in Health and Sport, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUC_2024_36
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Therapy Protocol (Other): Protocol for manual intervention using manual techniques on musculoskeletal structures
  Interventions: Other: Manual Therapy Protocol
- Sham Manual Protocol (Other): Manual sham intervention protocol through the application of manual contacts on musculoskeletal structures similar to the experimental group but without similar intention or pressure
  Interventions: Other: Sham Protocol
- Control (Other): No manual intervention
  Interventions: Other: Control-no treatment

INTERVENTIONS:
Other: Manual Therapy Protocol — The techniques were divided into three main groups: first, those carried out in cervical, thoracic and upper limbs; second, lumbar, pelvic and lower limbs; and finally, only spine. The techniques are carried out by physiotherapists with more than 15 years of healthcare experience and trained in manual therapy with more than 10 years of experience in this field.
  Arms: Manual Therapy Protocol
Other: Sham Protocol — The placebo protocol places the hands on the same areas as the experimental one and for the same application time but without making a manipulative intervention.
  Arms: Sham Manual Protocol
Other: Control-no treatment — Control group without treatment or manual contact
  Arms: Control

SUMMARY:
The study aims to observe the influence of manual therapy on physical and sporting performance. Manual therapy and physiotherapy have always been associated with post-exercise or as a means of recovering from injuries. The objective is to see if a physiotherapy intervention based on manual therapy causes changes in physical and sporting performance.

To do this, after a brief warm-up, a series of sports tests will be carried out, where the investigators will measure variables such as strength, range of motion, and autonomic nervous system parameters. Subsequently, a series of techniques will be applied in various anatomical regions, and finally, the sports tests will be repeated, and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Engage in low- or moderate-intensity physical activity.
* Engage in physical activity on 3 or more days per week.
* Not have any recent injury in the area of intervention that contraindicates manual intervention.
* Be willing to collaborate in the study.

Exclusion Criteria:

* Those people who had an acute injury or one that would prevent them from carrying out physical activity had any contraindication to the application of manual techniques.
* Who were not available during the dates of the study and people.
* Who were undergoing treatment with drugs that could interfere with the tests.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mobility | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  Measure joint mobility of the spine and upper and lower limbs through photo and video capture and subsequent evaluation with software. Measurements are also taken with goniometry and an inclinometer (angles and/or degrees).

SECONDARY OUTCOMES:
Strength | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  Measure the force (kilograms) of the column, lower and upper limbs through dynamometry capture, horizontal force in a treadmill, viewing the force in the Russian belt and jump test.
Speed | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  Measure the speed (metres/second) of the column, lower and upper limbs through jump, encoder, and race tests.
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  These parameters were evaluated before, during, and after the manual protocols were applied. For this purpose, the Elite HRV smartphone application was used, which connects to a Polar transmitter band placed on the person's chest at the level of the xiphoid process of the sternum, which allowed constant monitoring of the subject during each of the interventions.
  1. HRV analysis in time domain - SDNN (Standard Deviation of NN intervals): represents overall HRV and total autonomic activity. Units: ms.
  2. HRV analysis in time domain - RMSSD (Root Mean Square of Successive Differences): reflects parasympathetic (vagal) activity. Units: ms.
  3. HRV analysis in time domain - NN50 / pNN50 (Number or percentage of consecutive NN intervals differing by >50 ms): indicates short-term vagal regulation. Units: %.
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  These parameters were evaluated before, during, and after the manual protocols were applied. For this purpose, the Elite HRV smartphone application was used, which connects to a Polar transmitter band placed on the person's chest at the level of the xiphoid process of the sternum, which allowed constant monitoring of the subject during each of the interventions.
  1. HRV analysis in Frequency-Domain - Total Power (0-0.4 Hz): Overall HRV across all frequency bands. Units: ms².
  2. HRV analysis in Frequency-Domain - HF (High Frequency, 0.15-0.4 Hz): Reflects parasympathetic activity (vagal tone). Units: ms².
  3. HRV analysis in Frequency-Domain - LF (Low Frequency, 0.04-0.15 Hz): Represents sympathetic and parasympathetic activity. Units: ms².
  4. HRV analysis in Frequency-Domain LF/HF Ratio: Balance between sympathetic and parasympathetic activity. Units: ms².
Stress Salivary Test | Baseline; previous the first manual intervention and inmediatly posterior the first manual intervention (first day); 3, 7 and 14 days after the first manual intervention
  The Saliva Stress Test is a non-invasive diagnostic test that measures the levels of key stress biomarkers in the body's response. This analysis uses saliva samples collected at different times of the day (or night) to assess the rhythm of these biomarkers and their fluctuation.
  The saliva samples will be analysed for cortisol and IgA concentration using Ipro LFDs on a standard reader. After sample collection and mixing (2 minutes), two drops of saliva/buffer mix from the OFC will be added to the sample window of the cortisol or IgA LFFD.
  1. Cortisol measure. Unit: nM.
  2. IgA measure. Unit: µg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias de la Salud, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain